## Sleep-Disordered Breathing in the Acute Phase after Stroke and Neuropsychiatric Outcomes

2025-01-31

# Sleep-Disordered Breathing in the Acute Phase after Stroke and Neuropsychiatric Outcomes

### **Background/Objectives**

Stroke is the second leading cause of death and a common cause of acquired disability worldwide, and the burden of the disease at the societal level is expected to increase in the coming decades (1-4). Stroke can result in various long-term consequences, both neurological (such as aphasia, paresis, sensory or visual disturbances, and coordination and balance disorders) and neuropsychiatric (such as cognitive impairment, depression, and fatigue) (5-8). These consequences, in turn, affect stroke survivors' physical functions, activity levels, and ability to participate in daily activities (9-13).

Post-stroke fatigue is common, with prevalence estimates ranging between 25-85%, and 40% of stroke survivors have reported it as one of their worst symptoms (14-16). Recent Swedish studies have estimated the long-term prevalence 3-5 years after stroke to be between 24-52% (17, 18). Post-stroke fatigue partially overlaps with post-stroke depression, but approximately 70% of individuals with significant fatigue do not exhibit concurrent depressive symptoms (17). The condition is associated with poorer performance in daily activities and lower health-related quality of life (17). Currently, there are no specific treatments for post-stroke fatigue (19). Due to its high prevalence and consequences, it has recently been identified as one of the top ten priority research questions in stroke rehabilitation by the UK National Institute for Health and Care Research (20).

There are conflicting reports on whether traditional vascular risk factors such as hypertension, hyperlipidemia, heart disease (including atrial fibrillation), and smoking contribute to post-stroke fatigue (21, 22). Obesity is associated with post-stroke fatigue, and sleep-disordered breathing (SDB) has also emerged as a potential risk factor (23). Sleep-disordered breathing is prevalent after stroke, occurring in 50-70% of some populations (25). The dominant condition is obstructive sleep apnea syndrome (OSAS), followed by central sleep apnea (26). Established treatments for OSAS include continuous positive airway pressure (CPAP), mandibular advancement devices, surgical interventions, and weight loss (26), which can reduce daytime sleepiness. Research is ongoing regarding the extent to which treated OSAS can contribute to secondary prevention in stroke (27). Current American guidelines for secondary prevention provide a class 2b recommendation with moderate evidence for considering OSAS screening after stroke or transient ischemic attack (TIA) (28). The diagnosis is primarily made through overnight respiratory monitoring, with polysomnography being the gold standard, although it is time- and resource-intensive and may be cumbersome for the patient (29). Limited polygraphic examinations can also be conducted both in hospitals and at home (29).

#### **Research Questions:**

- 1. What is the 1-year prevalence of post-stroke fatigue in a hospital-based cohort in Blekinge?
- 2. How many individuals with stroke have significant sleep-disordered breathing according to non-invasive measurement?
- 3. What proportion of individuals with post-stroke fatigue had significant sleep-disordered breathing during hospitalization?
- 4. Can early, non-invasive, and simple measurement of sleep-disordered breathing in hospitals predict a subgroup of stroke patients who will develop significant fatigue?
- 5. Is there evidence that treatment goals after stroke are achieved to a lesser extent in those with significant fatigue?

By answering these questions, our study aims to: i) Facilitate patient selection for potential future clinical trials, e.g., CPAP treatment for preventing/treating post-stroke fatigue. ii) Identify potential subgroups among individuals with post-stroke fatigue. iii) Investigate risk factors for post-stroke fatigue, including sleep-disordered breathing. iv) Examine whether fatigue leads to poorer adherence to secondary preventive treatment goals (30).

#### Methodology

The present study has been approved by the Swedish Ethical Review Authority, diary number 2024-02659-01.

Study participants will be prospectively identified at the Department of Medicine, Blekinge Hospital, Karlskrona. Inclusion and exclusion criteria are as follows:

#### Inclusion criteria:

- Age >18 years
- Stroke according to WHO definition (31) (ischemic stroke, intracerebral hemorrhage, or subarachnoid hemorrhage)
- TIA with MRI-verified lesions corresponding to symptoms
- Informed consent to participate

#### Exclusion criteria:

- Traumatic stroke
- Tumor-associated bleeding
- Expected survival <3 months
- Unconsciousness (RLS >3)

Potential participants will be identified by medical staff, and informed consent will be obtained by a researcher.

Upon obtaining consent, patients will be equipped with a Withings Sleep Analyzer and a Nonin WristPro 2 pulse oximeter during hospital stay days 1- 3. Withings Sleep Analyzer is validated to detect moderate-severe obstructive sleep apnea (32). The patient is also equipped with a Nonin WristPro 2 pulse oximeter with the possibility to retrospectively obtain registered data regarding nocturnal hypoxia (T90 – time under 90% oxygen saturation, and ODI – oxygen desaturation index).

Baseline data collected include:

- National Institutes of Health Stroke Scale (NIHSS) (33)
- Pre-stroke modified Rankin Scale (mRS) (34)
- Previous stroke history
- BMI
- STOP-BANG questionnaire (35)

If it is not possible to obtain these data, including NIHSS, during the hospital stay, they will be collected later through chart review when possible. During chart review/clinical examination, the following will also be recorded:

- Main subtype of stroke (IS, ICH, SAH)
- Oxfordshire Community Stroke Project classification (OCSP) (36)
- Trial of Org 10172 in acute stroke treatment (TOAST) classification (37)
- Charlson Comorbidity Index (CCI) (38)
- Hypertension (>140/90 mmHg at discharge or antihypertensive treatment in the last 2 weeks)
- Diabetes mellitus (previous diagnosis, fasting blood glucose >6.1 mmol/L, or non-fasting blood glucose >11 mmol/L)
- Heart disease (ischemic heart disease, previous MI, angina, PCI, CABG, heart failure, arrhythmias)
- Hyperlipidemia (previous diagnosis, lipid-lowering treatment, total cholesterol >5 mmol/L, LDL >3 mmol/L)
- Smoking
- COPD (ICD-10 J44 or described in chart)
- Depression diagnosis (ICD F32-33) or antidepressant treatment
- HbA1c, lipid status, blood pressure at discharge
- Medications (antiplatelets, anticoagulants, antidiabetics, antihypertensives, opioids, sedatives, statins, antidepressants) at onset and discharge
- Long-term ECG monitoring
- Carotid stenosis degree on carotid ultrasound exam
- Coagulation assessment, if performed
- Previous stroke/recurrent stroke within 1 year

Participants are subsequently invited via letter for a follow-up visit approximately 1 year after stroke (+3 months, but not earlier than 1 year) at the district nurse students' training clinic at Blekinge Institute of Technology. During this visit, the following will be recorded: Follow-up assessment (1 year after stroke):

- Fatigue Assessment Scale (FAS) (39)
- Fatigue Visual Analogue Scale (VAFS)
- PHQ-9 depression scale (40)
- mRS (34)
- Blood pressure
- Height, weight, BMI
- Blood tests (HbA1c, lipid profile)
- Smoking
- Medication adherence
- Stroke Impact Scale (41)
- Ongoing BiPAP or CPAP treatment
- Alcohol consumption

#### **Recruitment Calculation**

With a confidence level of 0.05, statistical power of 80%, an estimated OSAS prevalence of 50%, and estimated significant fatigue prevalence of 30%, a total cohort of 284 participants is required to detect a doubled relative risk of significant fatigue with OSA. Considering a 10-20% loss to follow-up, approximately 340 participants need to be included.

#### **Ethical Considerations**

The project involves non-invasive procedures except for blood sampling at follow-up. Written informed consent will be obtained.

Data for research purposes such as apnea-hypopnea index and time under 90% blood oxygen saturation are collected outside of clinical praxis and do not in any way hinder concurrent investigation for OSA if clinically indicated. The sleep study data will be interpreted at the 1-year follow-up and the study physicians will decide if further investigation is needed.

#### **Affiliated Researchers**

Researcher Joseph Aked is the principal investigator, with Anders Behrens and Arne Lindgren as co-investigators.

#### References

- 1. GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019 Lancet. 2020;396:1204-1222. doi:10.1016/S0140-6736(20)30925-9.
- 2. GBD 2016 DALYs and HALE Collaborators: Global, regional, and national disability-adjusted life-years (DALYs) for 333 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990–2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet 2017; 390: 1260–1344.
- 3. Feigin VL, Krishnamurthi RV, Parmar P, Norrving B, et al: Update on the global burden of ischemic and hemorrhagic stroke in 1990–2013: the GBD 2013 Study. Neuroepidemiology 2015;45:161–176
- 4. Wafa HA, Wolfe CDA, Emmett E, et al. Burden of Stroke in Europe: Thirty- Year Projections of Incidence, Prevalence, Deaths, and Disability-Adjusted Life Years. Stroke 2020;51:2418-2427. doi: 10.1161/STROKEAHA.120.029606. Epub 2020 Jul 10. PMID: 32646325; PMCID: PMC7382540.
- 5. Feigin VL, Barker-Collo S, Parag V, et al. Auckland Stroke Outcomes Study. Part 1: Gender, stroke types, ethnicity, and functional outcomes 5 years poststroke. Neurology 2010;75:1597-1607.
- 6. Barker-Collo S, Feigin VL, Parag V, et al. Auckland Stroke Outcomes Study. Part 2: Cognition and functional outcomes 5 years poststroke. Neurology 2010;75:1608-1616
- 7. Jönsson AC, Delavaran H, Iwarsson S, et al. Functional status and patient-reported outcome 10 years after stroke: the Lund Stroke Register. Stroke 2014;45:1784-1790.
- 8. Cumming TB, Packer M, Kramer SF, et al. The prevalence of fatigue after stroke: A systematic review and meta-analysis. Int J Stroke 2016;11:968-977. doi:10.1177/1747493016669861.
- 9. Delavaran H, Jönsson AC, Lövkvist H, et al. Cognitive function in stroke survivors: A 10-year follow-up study. Acta Neurol Scand 2017;136:187-194. doi:10.1111/ane.12709
- 10. Stolwyk RJ, Mihaljcic T, Wong DK, et al. Poststroke Cognitive Impairment Negatively Impacts Activity and Participation Outcomes: A Systematic Review and Meta-Analysis. Stroke 2021;52:748-760. doi:10.1161/STROKEAHA.120.032215 11. Ayerbe L, Ayis S, Crichton S, et al. The natural history of depression up to 15 years after stroke: the South London Stroke Register. Stroke 2013;44:1105–1110. doi:
- 10.1161/STROKEAHA.111.679340
- 12. Christensen D, Johnsen SP, Watt T, et al. Dimensions of post-stroke fatigue: a two-year follow-up study. Cerebrovasc Dis 2008;26:134–141. doi: 10.1159/00013966
- 13. van de Port IGL, Kwakkel G, Schepers VPM, et al. Is fatigue an independent factor associated with activities of daily living, instrumental activities of daily living and health-related quality of life in chronic stroke? Cerebrovasc Dis 2007;23:40–45.
- 14. Cumming TB, Packer M, Kramer SF, et al. The prevalence of fatigue after stroke: A systematic review and meta-analysis. Int J Stroke 2016;11:968-977. doi:10.1177/1747493016669861
- 15. Elf M, Eriksson G, Johansson S, von Koch L, Ytterberg C (2016) Self-Reported Fatigue and Associated Factors Six Years after Stroke. PLOS ONE 11(8): e0161942. https://doi.org/10.1371/journal.pone.0161942
- 16. Pedersen A, Almkvist E, Holmegaard L, Lagging C, Redfors P, Blomstrand C, Jood K et al (2022) Fatigue 7 years post-stroke: Predictors and correlated features. Acta Neurol Scand. https://doi.org/10.1111/ane.13665
- 17. Aked J, Delavaran H, Wennerström F, et al. Cognition, fatigue and depression up to four years after first-ever stroke. Unpublished manuscript (2023).

- 18. Schnitzer, L., Hansson, PO., Samuelsson, C.M. et al. Fatigue in stroke survivors: a 5-year follow-up of the Fall study of Gothenburg. J Neurol (2023). https://doi.org/10.1007/s00415-023-11812-0
- 19. Wu S, Kutlubaev MA, Chun HYY, et al. Interventions for post-stroke fatigue. Cochrane Database Syst Rev. 2015;CD007030
- 20. Stroke rehabilitation and long-term care top 10 priorities.
- https://www.jla.nihr.ac.uk/priority-setting-partnerships/Stroke/stroke-rehabilitation-and-long term-care-top-10-priorities.htm. Accessed 4 Oct 2023.
- 21. Pedersen A, Almkvist E, Holmegaard L, Lagging C, Redfors P, Blomstrand C, Jood K et al (2022) Fatigue 7 years post-stroke: Predictors and correlated features. Acta Neurol Scand. https://doi.org/10.1111/ane.13665
- 22. Mahon S, Parmar P, Barker-Collo S, Krishnamurthi R, Jones K, Theadom A, Feigin V (2017) Determinants, prevalence, and trajectory of long-term post-stroke cognitive impairment: results from a 4-year follow-up of the ARCOS-IV study. Neuroepidemiology 3–4:129–134
- 23. Gu M, Xiao L, Wang J, Cai Q, Liu Y, Xu P, Liu Y et al (2021) Obesity and poststroke fatigue: a 2-year longitudinal study. Neurol Ther 2:955–969. https://doi.org/10.1007/s40120-021-00276-x
- 24. Kuvat N, Tanriverdi H, Armutcu F (2020) The relationship between obstructive sleep apnea syndrome and obesity: a new perspective on the pathogenesis in terms of organ crosstalk. Clin Respir J 7:595–604. https://doi.org/10.1111/crj.13175
- 25. Seiler A, Camilo M, Korostovtseva L, Haynes AG, Brill AK, Horvath T, Egger M, Bassetti CL. Prevalence of sleep-disordered breathing after stroke and TIA: a meta-analysis..Neurology. 2019; 92:e648–e654. doi: 10.1212/WNL.00000000000000904
- 26. Stevens D, Tomazini Martins R, Mukherjee S, et al. Post-stroke sleep-disordered breathing pathophysiology and therapy options. Front Surg. 2018;5:9
- 27. Boulos MI, Dharmakulaseelan L, Brown DL, et al. Trials in Sleep Apnea and Stroke. Stroke. 2021;51:366-372
- 28. Kleindorfer DO, Towfighi A, Chaturvedi S, et al. 2021 Guideline for the Prevention of Stroke in Patients with Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021;52:e364-e467
- 29. Hedner J GL, Friberg D, Ejnell H, Harlid R, Isacsson G, Lindberg E, Midgren B, Puzio J, Tegelberg Å, Ulander M, Wartenberg C. Riktlinjer för utredning av misstänkt sömnapné hos vuxna. Nationellt Kvalitetsregister SESAR/Registercentrum Väst; 2018. 1-39
- 30. Socialstyrelsen, Nationella riktlinjer för vård vid stroke 2018 Nationella riktlinjer för vård vid stroke Socialstyrelsen
- 31. Sacco RL, Kasner SE, Broderick JP, et al. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke 2013;44:2064-2089. doi:10.1161/STR.0b013e318296aeca.
- 32. Edouard P, Campo D, Bartet P, et al. Validation of the Withings Sleep Analyzer, an under-the-mattress device for the detection of moderate-severe sleep apnea syndrome. J Clin Sleep Med. 2021;17;1217-1227
- 33. Lyden P. Using the National Institutes of Health Stroke Scale: A Cautionary Tale. Stroke. 2017 Feb;48(2):513-519. doi: 10.1161/STROKEAHA.116.015434. Epub 2017 Jan 11. PMID: 28077454.
- 34. Bamford, J. M., Sandercock, A. G., Warlow, C. P., Slattery, J. (1989). Interobserver agreement for the assessment of handicap in stroke patients (letter). Stroke, 20, 828.
- 35. Hwang, M., Zhang, K., Nagappa, M., Saripella, A., Englesakis, M., & Chung, F. (2021). Validation of the STOP-Bang questionnaire as a screening tool for obstructive sleep apnoea

in patients with cardiovascular risk factors: a systematic review and meta-analysis. BMJ open respiratory research. 8(1), e000848. https://doi.org/10.1136/bmjresp-2020-000848

- 36. Bamford J, Sandercock P, Dennis M, et al. Classification and natural history of clinically identifiable subtypes of cerebral infarction. Lancet. 1991;337:1521-1526.
- 37. Adams HP, Bendixen BH, Kappelle LJ, et al. Classification of subtype of acute ischemic stroke: definitions for use in a multicenter clinical trial. Stroke. 1993;24:35-41
- 38. Hude Q, Bing L, Chantal MC, et al. Updating and Validating the Charlson Comorbidity Index and Score for Risk Adjustment in Hospital Discharge Abstracts Using Data From 6 Countries. American Journal of Epidemiology. 2011;173:676-682.
- 39. Cumming TB, Mead G. Classifying post-stroke fatigue: Optimal cut-off on the Fatigue Assessment Scale. Journal of Psychosomatic Research. 2017;103:147-149
- 40. Williams LS., Brizendine J, Plue L, et al. Performance of the PHQ-9 as a screening tool for depression after stroke. Journal of the American Heart Association. 2005;36:635-638
- 41. Duncan PW, Wallace D, Lai SM, et al. The Stroke Impact Scale version 2.0: Evaluation of reliability, validity, and sensitivity to change. Stroke 1999;30:2131-2140